CLINICAL TRIAL: NCT00569543
Title: Effects of Therapeutic Agents on Estrogens in the Breast
Brief Title: Effect of Tamoxifen or an Aromatase Inhibitor on Estrogen Metabolism in Women Treated for Newly Diagnosed Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0081-05-FB; P30CA036727 (NIH)
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: breast cancer in situ; ductal breast carcinoma in situ; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating | interventions — Chromatography, High Pressure Liquid; Mass Spectrometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: high performance liquid chromatography — urine analysis
Other: laboratory biomarker analysis — The biomarkers of interest will be the metabolites 4-OHE1(E2), estrogen-GSH conjugates and depurinating estrogen-DNA adducts.
Other: mass spectrometry — The urine samples will be analyzed for 40 estrogen metabolites, conjugates and depurinating DNA adducts by UPLC with tandem mass spectrometric detection.
Other: medical chart review — Collection of information about age, race, general health, any endocrine disorders, history of cancer, estrogen and progesterone receptor status, menopausal status and breast disease.

SUMMARY:
RATIONALE: Studying samples of urine in the laboratory from women with breast cancer may help doctors learn whether tamoxifen and aromatase inhibitors alter the metabolism of estrogens.

PURPOSE: This clinical trial is studying the effect of tamoxifen or an aromatase inhibitor on estrogen metabolism in women undergoing treatment for newly diagnosed breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Learn the effects of selected chemotherapy agents on the profile of estrogen metabolites, glutathione conjugates, and depurinating DNA adducts in urine from women with breast cancer.
* Determine whether tamoxifen citrate or aromatase inhibitor alters the metabolism of estrogens.

OUTLINE: Patients are stratified according to planned therapy (tamoxifen citrate vs aromatase inhibitor).

Patients receive tamoxifen citrate or an aromatase inhibitor as planned. Urine samples (and nipple aspirate fluid, if possible) are collected before beginning treatment and after 2-6 months of treatment. Samples are analyzed for 40 estrogen metabolites, conjugates, and depurinating DNA adducts by ultraperformance liquid chromatography with tandem mass spectrometric detection.

Patients' information, including race, body mass index, age at menarche, menopausal status, age at menopause if applicable, smoking history, alcohol consumption, pregnancy history including age at each pregnancy, lactation, history of benign breast disease, hysterectomy, and disease type, is collected through medical record review.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ductal carcinoma in situ or invasive breast cancer
* Scheduled to receive tamoxifen citrate or an aromatase inhibitor
* Estrogen receptor or progesterone receptor positive
* ECOG performance status 0, 1, or 2

Exclusion Criteria:

* Not pregnant or nursing
* No prior antiestrogen drug such as tamoxifen citrate or raloxifene
* No concurrent estrogens

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women newly diagnosed with breast cancer that will be given tamoxifen or an aromatase inhibitor for therapeutic reasons.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2005-05-11 (Actual); Primary Completion 2012-08-02 (Actual); Study Completion 2012-08-02 (Actual)

PRIMARY OUTCOMES:
Comparison of estrogen compounds in urine | before and after treatment for two-to-six months
  Comparison of estrogen compounds in urine before and after treatment with tamoxifen or an aromatase inhibitor for two-to-six months

CONTACTS AND LOCATIONS:
Overall Officials: Ercole Cavalieri, DSc, Principal Investigator — Eppley Cancer Center at University of Nebraska Medical Center
Locations (2):
- United States (2):
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Eppley Cancer Center at University of Nebraska Medical Center, Omaha, Nebraska